CLINICAL TRIAL: NCT05887973
Title: Addressing Root Causes for Gun Violence Prevention (ARC-GVP) Outcomes Study
Brief Title: Addressing Root Causes for Gun Violence Prevention (ARC-GVP)
Status: Recruiting | Type: Observational
Sponsor: University of Michigan (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Principal Investigator, Marc A. Zimmerman, Principal Investigator, University of Michigan
Other Study IDs: HUM00215637
Record Dates: First submitted 2023-03-30; First posted 2023-06-05 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Violence; Adolescent; Firearm Injury; Aggression
Keywords: Youth Violence Prevention; Gun Violence Prevention; Positive Youth Development
MeSH Terms: conditions — Aggression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Wave 1: Youth participants who are enrolled in The T.R.I.G.G.E.R Project's summer youth employment program in 2022
  Interventions: Behavioral: The T.R.I.G.G.E.R Project
- Wave 2: Youth participants who are enrolled in The T.R.I.G.G.E.R Project's summer youth employment program in 2023
  Interventions: Behavioral: The T.R.I.G.G.E.R Project
- Wave 3: Youth participants who are enrolled in The T.R.I.G.G.E.R Project's summer youth employment program in 2024
  Interventions: Behavioral: The T.R.I.G.G.E.R Project
- Wave 4: Youth participants who are enrolled in The T.R.I.G.G.E.R Project's summer youth employment program in 2025
  Interventions: Behavioral: The T.R.I.G.G.E.R Project

INTERVENTIONS:
Behavioral: The T.R.I.G.G.E.R Project — The T.R.I.G.G.E.R Project includes the following core components to address root causes of gun violence:
  * Summer Employment
  * Social and Emotional Learning
  * Future Orientation
  * Adult and Peer Support
  * Critical Consciousness
  * Civic Efficacy and Engagement

SUMMARY:
The goal of this study is to help build the evidence base for a locally-relevant youth firearm violence prevention program in Washington D.C., a city experiencing disparities in youth firearm violence outcomes.

The main question it aims to answer is:

How is youth participation in the summer youth employment program, the True Reasons I Grabbed the Gun Evolved from Risk (The T.R.I.G.G.E.R Project), which is designed to address root causes of gun violence, associated with individual youth behavioral outcomes, including pro-social involvement, aggression, and firearm-related attitudes and behaviors?

DETAILED DESCRIPTION:
The goal of this study is to help build the evidence base for a locally-relevant youth firearm violence prevention program in a city experiencing disparities in youth firearm violence outcomes. The main question it aims to answer is:

How is youth participation in a summer youth employment program that is designed to address root causes of gun violence (The T.R.I.G.G.E.R project), associated with individual youth behavioral outcomes, including pro-social involvement, retaliatory attitudes, aggression, and firearm behaviors?

To examine this question, participants will be invited to complete four surveys over the course of one year to assess attitudinal and behavioral change:

* A pre-test at the start of the program
* A first post-test 2-4 weeks following the conclusion of the program
* A second post-test 6 months following the conclusion of the program
* A third and final post-test 12 months following the conclusion of the program

ELIGIBILITY:
Inclusion Criteria:

* Youth in Washington D.C. who are participating in The T.R.I.G.G.E.R Project, a grassroots youth firearm violence prevention program

Exclusion Criteria:

* Emancipated minors

Ages: 14 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Youth in Washington D.C. who are participating in The T.R.I.G.G.E.R Project, a grassroots youth firearm violence prevention program
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2022-06-27 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Change in Civic Efficacy | Outcomes will be measured at 4 time points over 1 year: at the start of the summer programs, 2-4 weeks post, 6-months post, and 1-year post participation
  The investigators will assess change in civic efficacy (i.e., youth participants' sense of belief that they can create positive change in their communities) over time using the 3-item Civic Efficacy scale; the unit(s) of measurement are the Mean and Standard Deviation of scale scores; Minimum Value: 1 Maximum Value: 5, higher scores indicate a better outcome
Change in Pro-Social Involvement | Outcomes will be measured at 4 time points over 1 year: at the start of the summer programs, 2-4 weeks post, 6-months post, and 1-year post participation
  The investigators will assess change in pro-social involvement (i.e., youth participants' involvement in pro-social community organizations and activities) over time using an 8-item adapted Participation in Groups and Voluntary Organizations scale; the units of measurement are the Mean and Standard Deviation of scale scores; Minimum Value: 0 Maximum Value: 8; higher scores indicate a better outcome
Change in Attitudes towards Violence and Retaliation | Outcomes will be measured at 4 time points over 1 year: at the start of the summer programs, 2-4 weeks post, 6-months post, and 1-year post participation
  The investigators will assess change in youth participants' attitudes toward violence and retaliation over time using a 3-item Retaliatory Attitudes scale; the units of measurement are the Mean and Standard Deviation of scale scores; Minimum Value: 1 Maximum Value: 5; lower scores indicate a better outcome
Change in Aggressive Behavior | Outcomes will be measured at 4 time points over 1 year: at the start of the summer programs, 2-4 weeks post, 6-months post, and 1-year post participation
  The investigators will assess change in non-firearm related aggressive behavior (i.e., fighting, non-firearm weapon carriage) over time using a 3-item Aggressive Behaviors scale; the unit(s) of measurement are the Mean and Standard Deviation of scale scores; Minimum: 0, Maximum: 15, lower scores indicate a better outcome
Change in Firearm Carriage Frequency | Outcomes will be measured at 4 time points over 1 year: at the start of the summer programs, 2-4 weeks post, 6-months post, and 1-year post participation
  The investigators will assess change in the frequency of firearm carriage (for any reason besides hunting, target shooting, competitive shooting, or recreation) over time using 1-item; the unit(s) of measurement are the Mean and Standard Deviation of scale scores; Minimum: 1 Maximum: 7, lower scores indicate a better outcome
Change in Firearm Use | Outcomes will be measured at 4 time points over 1 year: at the start of the summer programs, 2-4 weeks post, 6-months post, and 1-year post participation
  The investigators will assess change in youth participants' firearm use (i.e., handling a gun, firing a gun, holding a gun in a selfie) over time, using a three-item Firearm Use scale; the unit(s) of measurement are the Means and Standard Deviations of scale scores, Minimum: 0 Maximum: 18, lower scores indicate a better outcome
Change in Firearm Aggression | Outcomes will be measured at 4 time points over 1 year: at the start of the summer programs, 2-4 weeks post, 6-months post, and 1-year post participation
  The investigators will assess change in youth participants' firearm aggression (i.e., threatening someone with a gun, firing at or around someone), using a two-item scale adapted from the Revised Conflict Tactics Scale; the unit(s) of measurement are the Means and Standard Deviations of scale scores, Minimum: 0 Maximum: 10, lower scores indicate a better outcome

CONTACTS AND LOCATIONS:
Overall Officials: Marc Zimmerman, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: Yes
The investigators will archive the data collected for this study in the Institute for Firearm Injury Prevention (IFIP) Data Repository so that the data will be connected to a national data resource on firearm injury prevention research. The IFIP repository is housed online at the Inter-University Consortium for Social and Political Research (ICPSR) (https://www.openicpsr.org/openicpsr/facts-open). All data uploaded to the repository will be de-identified, such that all sensitive, identifiable, or potentially identifiable information will be removed from the dataset. At a minimum, each data deposit in the archive will include the data set(s), codebook, data collection instrument, and a summary of the project.
Supporting Information: Study Protocol
Time Frame: All final data collected during the course of this research will be disseminated in a timely manner and as completely and accurately as possible, in accordance with Centers for Disease Control policy. The investigators will make the final version of the collected public health datasets available in a non-proprietary format within 30 months after the end of data collection in September 2026 via the Institute for Firearm Injury Prevention (IFIP) Data Repository portal. All identifiers will be removed from the data prior to dissemination. In compliance with the 1996 Health Insurance Portability and Accountability Act (HIPPA) wherever applicable. The data will be provided in standard file formats accompanied by the necessary documentation to allow for independent analyses. Once deposited, the de-identified data will be publicly available indefinitely.
Access Criteria: The de-identified data set(s) will be made publicly available without restrictions
URL: https://www.openicpsr.org/openicpsr/facts-open

REFERENCES:
- [Background] Crocetti E, Jahromi P, Meeus W. Identity and civic engagement in adolescence. J Adolesc. 2012 Jun;35(3):521-32. doi: 10.1016/j.adolescence.2011.08.003. Epub 2011 Aug 24. PMID 21868083
- [Background] Copeland-Linder N, Jones VC, Haynie DL, Simons-Morton BG, Wright JL, Cheng TL. Factors associated with retaliatory attitudes among African American adolescents who have been assaulted. J Pediatr Psychol. 2007 Aug;32(7):760-70. doi: 10.1093/jpepsy/jsm007. Epub 2007 Apr 2. PMID 17403911
- [Background] Black, S., & Hausman, A. (2008). Adolescents' views of guns in a high-violence community. Journal of Adolescent Research, 23(5), 592-610. http://doi.org/10.1177/0743558408322142
- [Background] Multisite Violence Prevention Project. The multisite violence prevention project: background and overview. Am J Prev Med. 2004 Jan;26(1 Suppl):3-11. doi: 10.1016/j.amepre.2003.09.017. PMID 14732182
- [Background] Straus, M., Hamby, S., Boney-McCoy, S., Sugarman, D. (1996). The Revised Conflict Tactics Scales (CTS2): Development and preliminary psychometric data. Journal of Family Issues, 17(3), 283-316.